CLINICAL TRIAL: NCT00894712
Title: Effect of Topical Application of Sulforaphane- Containing Broccoli Sprout Extracts on Radiation Dermatitis During External-beam Radiation Therapy for Breast Cancer
Brief Title: Topical Application of Sulforaphane-containing Broccoli Sprout Extracts on Radiation Dermatitis
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J-0838; NA_00018779
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Dermatitis
Keywords: Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms; Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Sulforaphane-containing broccoli sprout extracts (active agent) — Topical application, prepared with acetone, 280 nml daily, 3 times a week.
Device: Vehicle (inactive control) — Subjects will have measurements of skin erythema using a device called a chromometer

SUMMARY:
The investigators plan to investigate the protective effects of topical sulforaphane-containing broccoli-sprout extracts (BSE) on radiation-induced dermatitis in women undergoing external-beam radiation therapy for breast cancer. Topical sulforaphane induces phase 2 enzymes that are protective against oxidants, electrophiles, and inflammation (Talalay and Fahey, 2001) - all of which are generated by both ultraviolet and ionizing radiation. Previous work from the investigators' group demonstrated that sulforaphane treatment protects against ultraviolet radiation-induced erythema of human skin (IRB protocol NA_00004897; Talalay et al. 2007). This investigation will extend the investigators' previous work by employing ionizing rather than ultraviolet radiation.

The investigators propose a two part sequential protocol (Study A and Study B). Both studies will involve women with breast cancer who have undergone lumpectomy and are scheduled for adjuvant external beam radiation treatment. In study A, the investigators will validate their technique for measurement of skin erythema using a device called a chromometer; no active agent will be applied (up to 6 women). Study B will follow completion of Study A. Study B will involve the application of broccoli sprout extracts (BSE) or vehicle alone to determine if sulforaphane can reduce radiation-induced erythema (27 women). Four adjacent, 1.5-cm diameter areas-of-interest on the affected breast will be located by means of an adhesive vinyl template which can be accurately and repeatedly placed at the same position. Two of the four areas will be treated with BSE (active agent) and two with vehicle (inactive control). BSE will be applied on three days weekly throughout the 5-week period of whole breast radiation. Erythema will be noninvasively quantified by measuring the red-reflectance of the skin with a chromometer up to three times weekly throughout treatment. A total of 33 patients are to be enrolled.

The investigators' objective is to determine and quantify the effect of topical BSE on radiation-induced skin erythema. This study will employ standard, clinically-accepted radiation doses and techniques that are safe and well tolerated. The safety and tolerability of both oral and topical broccoli sprout preparations is well established; no safety concerns have been noted. (Shapiro et al. 2006; Dinkova-Kostova et al. 2007).

ELIGIBILITY:
Inclusion Criteria:

* Must have pathologically confirmed invasive adenocarcinoma or ductal carcinoma in situ of the breast.
* Patients must have undergone segmental mastectomy (i.e., lumpectomy).
* Patients must not have received prior radiation therapy to the breast.
* Patients must not have active local-regional disease prior to registration.
* Patients must not be pregnant because of the potential for fetal harm as a result of radiation treatment. Women of child-bearing age will be given a serum pregnancy test prior to study entry to ensure they are not pregnant. They will also be counseled on the importance of avoiding pregnancy and hormonal contraception while undergoing radiation therapy.
* Patients must not have a serious medical or psychiatric illness which prevents informed consent or compliance with treatment.
* All patients must be informed of the investigational nature of this study and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Visible skin pathology, excessive freckles, or skin blemishes in the test area.
* History of skin disease or hypersensitivity and repeated contact allergies.
* Sarcoma or squamous cell histology.
* Metastatic disease to the breast.
* Current tobacco use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2012-11-15 (Actual); Study Completion 2012-11-15 (Actual)

PRIMARY OUTCOMES:
Variance of the skin erythema measurements due to non-radiation effects. | Week 0 and Week 1 of radiation treatment
Absolute change in red reflectance of the skin. | before and after radiation

SECONDARY OUTCOMES:
Clinical grade of dermatitis (per NCI CTCAE v3.0 guidelines) for each region. | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zellars, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States